CLINICAL TRIAL: NCT00130949
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase II, Exploratory Evaluation of ALGRX 4975 in Subjects With Acute Lateral Epicondylitis
Brief Title: ALGRX 4975 in the Treatment of Tennis Elbow
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AlgoRx Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4975-2-005-2; Eudra CT No : 2004-001000-12
Record Dates: First submitted 2005-08-15; First posted 2005-08-17 (Estimated); Last update posted 2006-12-20 (Estimated); Status verified 2005-08

CONDITIONS: Tennis Elbow
Keywords: Acute lateral epicondylitis; Tennis elbow; Capsaicin
MeSH Terms: conditions — Tennis Elbow

INTERVENTIONS:
Drug: ALGRX 4975

SUMMARY:
Tennis elbow is a painful condition that results from repetitive arm movement with overuse of muscles, e.g. when playing tennis. A single injection of ALGRX 4975 has the potential to reduce pain for a period of weeks to months. This study will test the efficacy and safety of ALGRX 4975 in the treatment of patients with tennis elbow.

DETAILED DESCRIPTION:
Lateral epicondylitis (tennis elbow) is a painful condition that affects 4 to 7 adults per 1000 annually and tends to involve the subject's dominant side. It typically results from repetitive arm movement with over use of muscles leading to small tears in the tendons attaching muscles of the forearm to the epicondyles that may progress to tendonitis. Pain on or around the lateral epicondyle may radiate down the subject's arm. Gripping or extending the wrist often intensifies the pain.

More than 40 possible treatments have been proposed, reflecting a lack of consensus about optimal management. Non-steroidal anti-inflammatory drugs (NSAIDs) are commonly used to treat tennis elbow, but there are no trials to date that have compared them with other painkillers and one study found no clinically important benefit over placebo. Use of corticosteroid injections provides mixed results in relief of pain and at times insufficient evidence to support their use. Although complications associated with steroid injection are relatively uncommon, when a complication does occur, it can result in severe and disabling consequences for the subject. A small proportion of subjects fail to respond to only one injection of corticosteroid and some subjects who initially improved at four weeks had worse symptoms by six months.

This study has been designed to evaluate the safety and efficacy of a single soft tissue injection of ALGRX 4975 at a dose of 100 µg in comparison to placebo in subjects with acute LE.

ELIGIBILITY:
Inclusion Criteria:

* Acute lateral epicondylitis (LE) of less than 3 months duration (subjects with recurrent acute LE may be included).
* A screening and baseline severity of pain on resisted wrist dorsiflexion score of moderate or greater intensity.
* Lidocaine responsive.
* A systolic and diastolic blood pressure not greater than 140 and 95 mm Hg, respectively.

Exclusion Criteria:

* Any clinically significant form of joint disease, elbow trauma or neuromuscular disorder at the elbow, other than acute LE.
* Physiotherapy treatment within the preceding 2 weeks, prior to Visit 1.
* Any systemic or local corticosteroids within the preceding 3 months, except nasal or inhaled steroids at less than or equal to 1000 mcg/day.
* A medical condition other than LE that requires the use of a pain medication.
* A peripheral sensory or motor neuropathy involving the upper extremities.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2004-11; Study Completion 2005-11

PRIMARY OUTCOMES:
Pain induced by resisted wrist dorsiflexion 4 weeks after treatment

SECONDARY OUTCOMES:
Pain induced by resisted wrist dorsiflexion (other than 4 weeks)
Grip strength
Pain experienced during the grip strength test
Pain in elbow over previous 24 hours
Effect on work
Tenderness elicited by investigator or designee
Subjects' global impression of change
Secondary outcomes are evaluated at 1, 2, 4, 8 and 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Vasko, MD PhD, Principal Investigator — Ortopedicko-Traumatologicka Klinika, Kosice, Slovak Republic
Locations (1):
- Ortopedicko-Traumatologicka Klinika, Košice, Slovakia